CLINICAL TRIAL: NCT03603639
Title: A Multicenter, Double-Blind, Randomized, Cross-Over Study Evaluating Pharmacodynamic Activity of E2730 in Adult Subjects With Photosensitive Epilepsy
Brief Title: A Study to Evaluate the Pharmacodynamic Activity of E2730 in Adult Participants With Photosensitive Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to efficacy reasons.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2730-A001-201
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Photosensitive Epilepsy
Keywords: E2730; Epilepsy; Photosensitive; Seizures; PPR; Anti-epileptic
MeSH Terms: conditions — Epilepsy, Reflex; Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo, E2730 40 mg, E2730 120 mg (Experimental): Participants will receive a single dose of E2730-matched placebo, capsule, orally (Treatment A) in Treatment Period 1 followed by a single dose of E2730 40 mg, capsule, orally (Treatment B) in Treatment Period 2 followed by a single dose of E2730 120 mg, capsule, orally (Treatment C) in Treatment Period 3. A wash-out phase of at least 3-weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2730
- E2730 40 mg, E2730 120 mg, Placebo (Experimental): Participants will receive a single dose of E2730 40 mg, capsule, orally (Treatment B) in Treatment Period 1 followed by a single dose of E2730 120 mg, capsule, orally (Treatment C) in Treatment Period 2 followed by a single dose of E2730-matched placebo, capsule, orally (Treatment A) in Treatment Period 3. A wash-out phase of at least 3-weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2730
- E2730 120 mg, Placebo, E2730 40 mg (Experimental): Participants will receive a single dose of E2730 120 mg, capsule, orally (Treatment C) in Treatment Period 1 followed by a single dose of E2730-matched placebo, capsule, orally (Treatment A) in Treatment Period 2 followed by a single dose of E2730 40 mg, capsule, orally (Treatment B) in Treatment Period 3. A wash-out phase of at least 3-weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2730
- Placebo, E2730 120 mg, E2730 40 mg (Experimental): Participants will receive a single dose of E2730-matched placebo, capsule, orally (Treatment A) in Treatment Period 1 followed by a single dose of E2730 120 mg, capsule, orally (Treatment C) in Treatment Period 2 followed by a single dose of E2730 40 mg, capsule, orally (Treatment B) in Treatment Period 3. A wash-out phase of at least 3-weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2730
- E2730 40 mg, Placebo, E2730 120 mg (Experimental): Participants will receive a single dose of E2730 40 mg, capsule, orally (Treatment B) in Treatment Period 1 followed by a single dose of E2730-matched placebo, capsule, orally (Treatment A) in Treatment Period 2 followed by a single dose of E2730 120 mg, capsule, orally (Treatment C) in Treatment Period 3. A wash-out phase of at least 3-weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2730
- E2730 120 mg, E2730 40 mg, Placebo (Experimental): Participants will receive a single dose of E2730 120 mg, capsule, orally (Treatment C) in Treatment Period 1 followed by a single dose of E2730 40 mg, capsule, orally (Treatment B) in Treatment Period 2 followed by a single dose of E2730-matched placebo, capsule, orally (Treatment A) in Treatment Period 3. A wash-out phase of at least 3-weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2730

INTERVENTIONS:
Drug: Placebo — Participants will receive E2730-matched placebo capsule, orally.
Drug: E2730 — Participants will receive E2730 capsule, orally.

SUMMARY:
The primary purpose of the study is to assess the pharmacodynamic (PD) activity of E2730 as measured by suppression of epileptic photoparoxysmal response (PPR) in the participant's most sensitive eye condition in participants with photosensitive epilepsy.

DETAILED DESCRIPTION:
Adult participants with epilepsy will be enrolled in this study. This study will consist of 2 phases: Prerandomization and Randomization Phase.

The Prerandomization Phase will consist of a Screening Period (up to 3 weeks), during which each participant's study eligibility will be determined and baseline assessments will be conducted. The Randomization Phase will consist of 3 Treatment Periods with a single dose in each period (placebo, E2730 40 mg, or E2730 120 mg), each separated by a 3-week washout interval for a total of approximately 6 weeks, and a Follow-up Period (3 weeks after the last dose of study drug).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 60 years old at the time of informed consent.
2. A diagnosis and history of a PPR on EEG with or without a diagnosis of epilepsy.
3. Currently taking up to a maximum of 3 concomitant antiepileptic drugs (AEDs). If taking concomitant AED(s), the dose must have remained stable for at least 4 weeks prior to Screening.
4. A reproducible intermittent photic stimulation (IPS)-induced PPR on EEG of at least 3 points on a frequency assessment scale (SPR) in at least 1 eye condition on at least 3 of the EEGs performed at Screening.
5. A body mass index (BMI) between 18 to 35 kilogram per square meter (kg/m^2) and a total body weight greater than or equal to 45 kilograms (kg) at the time of Screening.

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 international units per liter [IU/L] or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
2. History of nonepileptic seizures (eg, metabolic, structural, or pseudoseizures) while on any antiepileptic medication(s).
3. History of status epilepticus while on any antiepileptic medication(s) within 2 years prior to Screening.
4. Ongoing or history of generalized tonic-clonic seizures within 6 months prior to Screening.
5. Previously developed or who experienced a clinical seizure during prior PPR assessment or Screening IPS procedure, respectively.
6. Use of AEDs that affect gama-aminobutyric acid (GABA) (GABAergic AEDs) (such as tiagabine, vigabatrin, gabapentin, pregabalin) within 3 months prior to Screening.
7. Multiple drug allergies or a severe drug reaction to AED(s), including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity reactions.
8. An active central nervous system (CNS) infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
9. Concomitant use of cannabinoids.
10. Inability to follow restriction on watching television, or use of any device with an animated screen (ie, computer, video games, tablets).
11. A history of prolonged QT syndrome or risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome), or the use of concomitant medications that prolonged the QT/corrected QT (QTc) interval; or prolonged QT/QTc interval (QTc greater than [>] 450 millisecond [msec]) demonstrated on electrocardiograms (ECG) at Screening or baseline (based on average of triplicate ECGs).
12. Any suicidal ideation with intent with or without a plan within 6 months before Screening or during Screening (ie, answering "Yes" to questions 4 or 5 on the suicidal ideation section of the Columbia-Suicide Severity Rating Scale [C-SSRS]).
13. Any lifetime suicidal behavior (per the suicidal behavior section of the C-SSRS).
14. Any psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years.
15. Frequent spontaneous background burst or current evidence of proconvulsive activity on EEG (eg, increase in spike-wave activity) at Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Eisai Inc.
Locations (5):
- United States (5):
  - Clinical Trials, Inc. and Arkansas Epilepsy Program, Little Rock, Arkansas
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Johns Hopkins University- School of Medicine, Baltimore, Maryland
  - Washington University Hospital, St Louis, Missouri
  - Unniversity of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 27 July 2018 to 14 February 2019.
Pre-assignment Details: A total of 8 participants were screened, of which 2 were screen failures and 6 were randomized to receive study treatment. The study was terminated due to lack of photoparoxysmal response (PPR).
Groups:
- Sequence 1: Placebo + E2730 40 mg + E2730 120 mg: Participants received, E2730-matched placebo (Treatment A) capsule, orally, once on Day 1 in Treatment Period 1, followed by E2730 40 milligram (mg) (Treatment B) capsule, orally, once on Day 1 in Treatment Period 2, followed by E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 3. A washout period of at least 3 weeks was maintained between all the treatment periods.
- Sequence 2: E2730 40 mg + E2730 120 mg + Placebo: Participants received, E2730 40 mg (Treatment B) capsule, orally, once on Day 1 in Treatment Period 1, followed by E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 2, followed by E2730-matched placebo (Treatment A) capsule, orally, once on Day 1 in Treatment Period 3. A washout period of at least 3 weeks was maintained between all the treatment periods.
- Sequence 3: E2730 120 mg + Placebo + E2730 40 mg: Participants received, E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 1, followed by E2730 -matched placebo (Treatment A) capsule, orally, once on Day 1 in Treatment Period 2, followed by E2730 40 mg (Treatment B) capsule, orally, once on Day 1 in Treatment Period 3. A washout period of at least 3 weeks was maintained between all the treatment periods.
- Sequence 4: Placebo + E2730 120 mg + E2730 40 mg: Participants received, E2730-matched placebo (Treatment A) capsule, orally, once on Day 1 in Treatment Period 1, followed by E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 2, followed by E2730 40 mg (Treatment B) capsule, orally, once on Day 1 in Treatment Period 3. A washout period of at least 3 weeks was maintained between all the treatment periods.
- Sequence 5: E2730 40 mg + Placebo + E2730 120 mg: Participants received, E2730 40 mg (Treatment B) capsule, once on Day 1 in Treatment Period 1, followed by E2730 -matched placebo (Treatment A) capsule, orally, once on Day 1 in Treatment Period 2, followed by E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 3. A washout period of at least 3 weeks was maintained between all the treatment periods.
- Sequence 6: E2730 120 mg + E2730 40 mg + Placebo: Participants received, E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 1, followed by E2730 40 mg (Treatment B) capsule, orally, once on Day 1 in Treatment Period 2, followed by E2730-matched placebo (Treatment A) capsule, orally, once on Day 1 in Treatment Period 3. A washout period of at least 3 weeks was maintained between all the treatment periods.
Period: Treatment Period 1 (Day 1)
Arm/Group | Sequence 1: Placebo + E2730 40 mg + E2730 120 mg | Sequence 2: E2730 40 mg + E2730 120 mg + Placebo | Sequence 3: E2730 120 mg + Placebo + E2730 40 mg | Sequence 4: Placebo + E2730 120 mg + E2730 40 mg | Sequence 5: E2730 40 mg + Placebo + E2730 120 mg | Sequence 6: E2730 120 mg + E2730 40 mg + Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 3 Weeks)
Arm/Group | Sequence 1: Placebo + E2730 40 mg + E2730 120 mg | Sequence 2: E2730 40 mg + E2730 120 mg + Placebo | Sequence 3: E2730 120 mg + Placebo + E2730 40 mg | Sequence 4: Placebo + E2730 120 mg + E2730 40 mg | Sequence 5: E2730 40 mg + Placebo + E2730 120 mg | Sequence 6: E2730 120 mg + E2730 40 mg + Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 1)
Arm/Group | Sequence 1: Placebo + E2730 40 mg + E2730 120 mg | Sequence 2: E2730 40 mg + E2730 120 mg + Placebo | Sequence 3: E2730 120 mg + Placebo + E2730 40 mg | Sequence 4: Placebo + E2730 120 mg + E2730 40 mg | Sequence 5: E2730 40 mg + Placebo + E2730 120 mg | Sequence 6: E2730 120 mg + E2730 40 mg + Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 3 Weeks)
Arm/Group | Sequence 1: Placebo + E2730 40 mg + E2730 120 mg | Sequence 2: E2730 40 mg + E2730 120 mg + Placebo | Sequence 3: E2730 120 mg + Placebo + E2730 40 mg | Sequence 4: Placebo + E2730 120 mg + E2730 40 mg | Sequence 5: E2730 40 mg + Placebo + E2730 120 mg | Sequence 6: E2730 120 mg + E2730 40 mg + Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 0 | 1 | 1
Period: Treatment Period 3 (Day 1)
Arm/Group | Sequence 1: Placebo + E2730 40 mg + E2730 120 mg | Sequence 2: E2730 40 mg + E2730 120 mg + Placebo | Sequence 3: E2730 120 mg + Placebo + E2730 40 mg | Sequence 4: Placebo + E2730 120 mg + E2730 40 mg | Sequence 5: E2730 40 mg + Placebo + E2730 120 mg | Sequence 6: E2730 120 mg + E2730 40 mg + Placebo
Started | 1 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- All Participants: Participants received E2730-matched placebo (Treatment A) or E2730 40 mg (Treatment B) or E2730 120 mg (Treatment C) capsule, orally, once on Day 1 in Treatment Period 1 to 3 as per assigned treatment sequence. A washout period of at least 3 weeks was maintained between all the treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.32)
Age, Customized [Count of Participants; unit: Participants]
  greater than or equal to (>=) 18 to less than (<) 40 | 5
  >= 40 to < 60 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Standard Photosensitivity Response (SPR) in the Most Sensitive Eye Condition at 8 Hours Post-dose on Day 1 of Each Treatment Period
Description: Photosensitivity described the presentation of an epileptiform electroencephalogram (EEG) response PPR from exposure to intermittent photic stimulation (IPS). SPR was a standardized derived measure of the range of frequencies of IPS that elicits epileptiform EEG responses in a participant. The participants were exposed to 14 different frequencies ranging from 2 to 60 flashes per second. The range was then assigned a number, representing the number of frequency steps, ranging from 0 to 14 between the lowest to the highest frequencies of IPS that elicits epileptiform activity by EEG. The lower scores represented better outcomes. Day 1 as per assigned treatment sequence in Treatment Period 1, 2, or 3. Mean change from baseline in the SPR most sensitive eye condition was the average of SPR scores assessed post study drug administration (Day 1 of Treatment Period 1, 2, or 3).
Time Frame: Baseline (30 minutes-2 hours) pre-dose and at 8 hours post-dose on Day 1 of each treatment period
Population: The pharmacodynamic (PD) analysis set included randomized participants who received at least 1 dose of study drug and had sufficient PD data to derive at least 1 PD parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment A: Placebo: Participants received, E2730-matched placebo capsule, orally, once on Day 1 as per assigned treatment sequence in Treatment Period 1, 2, or 3.
- Treatment B: E2730 40 mg: Participants received, E2730 40 mg capsule, orally, once on Day 1 as per assigned treatment sequence in Treatment Period 1, 2, or 3.
- Treatment C: E2730 120 mg: Participants received, E2730 120 mg capsule, orally, once on Day 1 as per assigned treatment sequence in Treatment Period 1, 2, or 3.
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
units on a scale
  Baseline | 7.80 (5.495) | 5.50 (6.137) | 9.00 (3.391)
  Change at 8 hour post-dose | -0.12 (1.677) | 0.65 (0.755) | 1.00 (2.839)
Statistical Analysis 1: Comparison: Treatment A: Placebo vs Treatment B: E2730 40 mg; The mixed effects model for the crossover part of the study will include treatment, period, and sequence as fixed effects, baseline (Predose) measurement as a covariate, and subject nested within sequence as a random effect; Test type: Superiority; LS Mean difference = 1.38, 90% CI 2-sided [-0.72 to 3.48]
Statistical Analysis 2: Comparison: Treatment A: Placebo vs Treatment C: E2730 120 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; LS Mean difference = 1.07, 90% CI 2-sided [-0.49 to 2.63]

2. Secondary Outcome: Mean Change From Baseline in SPR in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Opened) at 8 Hours Post-dose on Day 1 of Each Treatment Period
Description: Photosensitivity described the presentation of an epileptiform EEG response PPR from exposure to IPS. SPR was a standardized derived measure of the range of frequencies of IPS that elicits epileptiform EEG responses in a participant. IPS-EEG assessments determine the range of frequencies of IPS that elicited an epileptiform EEG response. Each IPS-EEG assessment was conducted in all 3 eye conditions (eye closure, eyes closed, and eyes open). The participants were exposed to 14 different frequencies ranging from 2 to 60 flashes per second. The range was then assigned a number, representing the number of frequency steps, ranging from 0 to 14. Lower scores represented better outcomes. Mean change from baseline in the SPR in each of the 3 eye conditions (Eye Closure, Eyes Closed, and Eyes Opened) was the average of SPR scores assessed post study drug administration (Day 1 of Treatment Period 1, 2, or 3).
Time Frame: Baseline (30 minutes-2 hours) pre-dose and at 8 hours post-dose on Day 1 of each treatment period
Population: The PD analysis set included randomized participants who received at least 1 dose of study drug and had sufficient PD data to derive at least 1 PD parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
units on a scale
  Eye Closure: At Baseline | 8.00 (6.000) | 5.75 (6.551) | 9.20 (3.114)
  Eye Closure: Change at 8 hours post-dose | 0.12 (1.579) | 0.65 (1.279) | 0.60 (2.054)
  Eyes Closed: At Baseline | 7.60 (5.225) | 5.25 (6.021) | 8.80 (3.114)
  Eyes Closed: Change at 8 hours post-dose | -0.24 (1.711) | 0.90 (1.149) | 0.92 (2.969)
  Eyes Open: At Baseline | 4.20 (5.762) | 4.75 (6.185) | 7.00 (2.646)
  Eyes Open: Change at 8 hours post-dose | 0.76 (1.846) | 0.05 (1.716) | 1.20 (2.874)
Statistical Analysis 1: Comparison: Treatment A: Placebo vs Treatment B: E2730 40 mg; In eye closure condition. The mixed effects model for the crossover part of the study will include treatment, period, and sequence as fixed effects, baseline (Predose) measurement as a covariate, and subject nested within sequence as a random effect; Test type: Superiority; LS Mean Difference = 0.39, 90% CI 2-sided [-0.75 to 1.54]
Statistical Analysis 2: Comparison: Treatment A: Placebo vs Treatment C: E2730 120 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; LS Mean Difference = 0.30, 90% CI 2-sided [-0.60 to 1.21]
Statistical Analysis 3: Comparison: Treatment A: Placebo vs Treatment B: E2730 40 mg; In eyes closed condition. The mixed effects model for the crossover part of the study will include treatment, period, and sequence as fixed effects, baseline (Predose) measurement as a covariate, and subject nested within sequence as a random effect; Test type: Superiority; LS Mean Difference = 1.62, 90% CI 2-sided [-1.16 to 4.39]
Statistical Analysis 4: Comparison: Treatment A: Placebo vs Treatment C: E2730 120 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; LS Mean Difference = 1.05, 90% CI 2-sided [-0.89 to 2.98]
Statistical Analysis 5: Comparison: Treatment A: Placebo vs Treatment B: E2730 40 mg; In eyes open condition. The mixed effects model for the crossover part of the study will include treatment, period, and sequence as fixed effects, baseline (Predose) measurement as a covariate, and subject nested within sequence as a random effect; Test type: Superiority; LS Mean Difference = 0.21, 90% CI 2-sided [-1.87 to 2.28]
Statistical Analysis 6: Comparison: Treatment A: Placebo vs Treatment C: E2730 120 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; LS Mean Difference = 1.27, 90% CI 2-sided [-0.57 to 3.11]

3. Secondary Outcome: Time to Onset of Mean Photosensitivity Response in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Open Condition) up to 8 Hours Post-dose on Day 1 of Each Treatment Period
Description: Time to onset of mean photosensitivity response in each of the 3 eye conditions (eye closure, eyes closed, and eyes open condition) was determined from mean change from baseline SPR data across participants. The onset of mean suppression was defined as the first time point at which the mean SPR across participants (not for each participant) was at least 3 units below the mean SPR at baseline. Photosensitivity response were essentially intermittent photic stimulation IPS assessments, is a form of visual stimulation, when the participants are flashed with light on their eyes intermittently at different hertz.
Time Frame: Baseline (30 minutes-2 hours) pre-dose up to 8 hours post-dose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Number; unit: hours
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
hours
  Eye Closure | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment.
  Eyes Closed | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment.
  Eyes Opened | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment.

4. Secondary Outcome: Duration of Mean Photosensitivity Response in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Open Condition) up to 8 Hours Post-dose on Day 1 of Each Treatment Period
Description: Duration of mean photosensitivity response in each of the 3 eye conditions (eye closure, eyes closed, and eyes open condition) was determined from mean change from baseline SPR data across participants. Duration of suppression was defined as the difference in hours between the onset of suppression and the end of suppression of photosensitivity across participants. The onset of mean suppression was defined as the first time point at which the mean SPR across participants (not for each participant) was at least 3 units below the mean SPR at baseline. The end of mean suppression was defined as the last time (second time) with two successive reductions in mean SPR of at least 3 units lower than the mean SPR at baseline. SPR was a standardized derived measure of range of frequencies of IPS that elicits epileptiform EEG responses in a participant. The range was then assigned a number, representing the number of frequency steps, ranging from 0 to 14. Lower scores represented better outcomes.
Time Frame: Baseline (30 minutes-2 hours) pre-dose up to 8 hours post-dose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Number; unit: hours
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
hours
  Eye Closure: Duration | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment.
  Eyes Closed: Duration | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment.
  Eyes Open: Duration | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment.

5. Secondary Outcome: Number of Participants With Complete Suppression, Partial Response, and no Response of SPR up to 8 Hours Post-dose on Day 1 of Each Treatment Period
Description: Complete suppression was defined as a SPR reduction to 0 over at least 1 time point for all three eye conditions. Partial response was defined as a reduction in SPR of at least 3 units from baseline for at least 3 time points, and no time points with at least 3 units of increase, in the most sensitive eye condition; without meeting the complete suppression definition. No response was defined as the response not meeting complete suppression or partial suppression definitions.
Time Frame: Baseline (30 minutes-2 hours) pre-dose up to 8 hours post-dose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
Participants
  Complete Suppression | 0 | 0 | 0
  Partial Response | 1 | 0 | 0
  No Response | 4 | 4 | 5

6. Secondary Outcome: Maximum Change From Baseline of Photosensitivity Response in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Open Condition) up to 8 Hours Post-dose on Day 1 of Each Treatment Period
Description: Maximum change from baseline of photosensitivity response in each of the 3 eye conditions (eye closure, eyes closed, and eyes open condition) across participants (not for each participant) were reported. Photosensitivity described the presentation of an epileptiform EEG response (PPR) from exposure to IPS. SPR was a standardized derived measure of the range of frequencies of IPS that elicits epileptiform EEG responses in a participant. IPS-EEG assessments determine the range of frequencies of IPS that elicited an epileptiform EEG response. Each IPS-EEG assessment was conducted in all 3 eye conditions (eye closure, eyes closed, and eyes open). The participants were exposed to 14 different frequencies ranging from 2 to 60 flashes per second. The range was then assigned a number, representing the number of frequency steps, ranging from 0 to 14. Lower scores representing better outcomes.
Time Frame: Baseline (30 minutes-2 hours) pre-dose up to 8 hours post-dose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Number; unit: units on a scale
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
units on a scale
  Eye Closure: Baseline | 14.0 | 14.0 | 13.0
  Eye Closure: Maximum change from baseline | 2.6 | 2.0 | 4.0
  Eyes Closed: Baseline | 13.0 | 13.0 | 12.0
  Eyes Closed: Maximum change from baseline | 1.6 | 2.4 | 6.0
  Eyes Open: Baseline | 11.0 | 13.0 | 10.0
  Eyes Open: Maximum change from baseline | 3.8 | 2.2 | 5.0

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAE was defined as an adverse event (AE) that emerged during treatment, having been absent at pretreatment (Baseline) or reemerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE is continuous. An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: First dose of study drug (Baseline) up to 28 days after last dose of study drug (Day 71)
Population: The safety analysis set included participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
Participants | 3 | 1 | 1

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline Values For Vital Signs
Description: Vital signs parameters included systolic and diastolic Blood Pressure, pulse rate, respiratory rate, and temperature were assessed. Clinically significant values were defined as values above or below the normal reference range post-dose. Number of participants with clinically significant change from baseline values for vital signs was reported.
Time Frame: First dose of study drug (Baseline) up to 28 days after last dose of study drug (Day 71)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline Values for Laboratory Parameters: Clinical Chemistry, Hematology and Liver Function Test
Description: Laboratory assessment included clinical chemistry, hematology and liver function test parameters. Clinically significant values were defined as values above or below the normal reference range post-dose. Number of participants with clinically significant change from baseline values for laboratory parameters: clinical chemistry, hematology and liver function test are reported.
Time Frame: First dose of study drug (Baseline) up to 28 days after last dose of study drug (Day 71)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
Participants
  Clinical Chemistry | 0 | 0 | 0
  Hematology | 0 | 0 | 0
  Liver Function Test | 0 | 0 | 0

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for E2730 and N-acetyl Metabolite
Time Frame: Days 1, 22 and 43: 0-8 hours post-dose
Population: The pharmacokinetic (PK) analysis set included randomized participants who received at least 1 dose of study drug and had sufficient PK data to derive at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 4 | 5
nanogram per milliliter (ng/mL)
  E2730 | 737 (18.4) | 2440 (18.5)
  N-acetyl metabolite | 0.672 (62.3) | 1.89 (38.2)

11. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration (Cmax) for E2730 and N-acetyl Metabolite
Time Frame: Days 1, 22 and 43: 0-8 hours post-dose
Population: The PK analysis set included randomized participants who received at least 1 dose of study drug and had sufficient PK data to derive at least 1 PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 4 | 5
hours
  E2730 | 4.15 [2.02 to 5.92] | 1.78 [0.10 to 7.93]
  N-acetyl metabolite | 1.65 [1.03 to 4.20] | 4.00 [0.10 to 7.93]

12. Secondary Outcome: AUC (0-8h): Area Under the Plasma Concentration-time Curve From 0 to 8 Hours Post-dose for E2730 and N-acetyl Metabolite
Time Frame: Days 1, 22 and 43: 0-8 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 4 | 5
hour*nanogram per milliliter (h*ng/mL)
  E2730 | 5140 (18.4) | 15100 (23.2)
  N-acetyl metabolite | 2.48 (183) | 10.0 (37.3)

13. Secondary Outcome: Model Based Relationship Between PK Parameters of E2730 and Onset, Maximum Change, and Duration of Impact on Photosensitivity
Description: Relationship between PK parameters of E2730 and PD parameters (onset, maximum change, and duration of impact on photosensitivity) were to be assessed using model-based approach. The PK-PD analysis dataset were to be used and included in examination of the relationship of PK of E2730 and change in PPR response (example, time of onset, maximum change, and duration of PPR; Bond and Lader data).
Time Frame: Baseline (30 minutes-2 hours) pre-dose up to 8 hours post-dose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
Number analyzed (Participants) | 5 | 4 | 5
correlation coefficient | NA — Relationship Between PK Parameters of E2730 and PD parameters (onset, maximum change, and duration of impact on photosensitivity) cannot be determined because no PPR and dose response was observed during assessment period. Hence, the PK-PD analysis was not conducted. | NA — Relationship Between PK Parameters of E2730 and PD parameters (onset, maximum change, and duration of impact on photosensitivity) cannot be determined because no PPR and dose response was observed during assessment period. Hence, the PK-PD analysis was not conducted. | NA — Relationship Between PK Parameters of E2730 and PD parameters (onset, maximum change, and duration of impact on photosensitivity) cannot be determined because no PPR and dose response was observed during assessment period. Hence, the PK-PD analysis was not conducted.

ADVERSE EVENTS:
Time Frame: Up to 28 days after last dose of study drug (Day 71)
Arm/Group | Treatment A: Placebo | Treatment B: E2730 40 mg | Treatment C: E2730 120 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 1/5
Other Adverse Events (participants affected / at risk) | 3/5 | 1/4 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Placebo (N=5) | Treatment B: E2730 40 mg (N=4) | Treatment C: E2730 120 mg (N=5)
Eyelid myoclonus (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Placebo (N=5) | Treatment B: E2730 40 mg (N=4) | Treatment C: E2730 120 mg (N=5)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT03603639/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03603639/SAP_001.pdf